CLINICAL TRIAL: NCT01780753
Title: A Study of the Pharmacokinetics of Primaquine in Lactating Women and Breastfed Infants for the Radical Treatment of Uncomplicated Maternal P. Vivax
Brief Title: Primaquine Pharmacokinetics in Lactating Women and Their Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMRU1203
Record Dates: First submitted 2012-10-08; First posted 2013-01-31 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Vivax Malaria
Keywords: Primaquine; Vivax malaria; G6PD
MeSH Terms: conditions — Malaria, Vivax | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Primaquine (Experimental): Primaquine GPO® (Government Pharmaceutical Organization, Thailand) 0.5 mg/kg will be given once daily for 14 days.
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: Primaquine — Primaquine GPO® (Government Pharmaceutical Organization, Thailand) 0.5 mg/kg will be given once daily for 14 days.

SUMMARY:
The weight of malaria falls most heavily on young children and pregnant women but studies of the safety of antimalarials in pregnancy and lactation are few. The only recommended medication used for radical treatment of P.vivax is primaquine. The 2010 WHO malaria guidelines recommend its use in all patients with P.vivax infection in areas of low transmission, in the absence of contraindications. Primaquine is contraindicated in pregnancy. The postpartum period presents a key opportunity to definitively treat women who suffer multiple malaria relapses during pregnancy. The 2010 WHO malaria treatment guidelines allow for primaquine use during lactation but there are no studies to date quantifying primaquine excretion in breast milk and the dose that breastfed infants would be exposed to is unknown. The investigators propose to study the pharmacokinetics of primaquine in maternal and infant plasma and in breast milk during a 14 day radical treatment of P.vivax.

Some inferences about the expected behavior of primaquine in lactation can be drawn from its known pharmacologic properties. Primaquine pharmacokinetics have been well characterized in healthy subjects and malaria patients after single and multiple oral dosing. Peak concentrations are reached within 2-3 hours after dosing and the plasma elimination half-life is ~7 hours. It is extensively distributed in the tissue and largely metabolized to inert carboxyprimaquine, the major plasma metabolite, which undergoes further biotransformation to unknown metabolites that are probably more toxic than the parent compound. The identification of other metabolites in humans has been difficult to pursue because the expected aminophenol metabolites are unstable.

No pharmacokinetic studies have been done to measure primaquine excretion in breast milk. A few studies have been done of other antimalarials during lactation and have shown low levels of drug in breast milk during treatment.

DETAILED DESCRIPTION:
Background The weight of malaria falls most heavily on young children and pregnant women but studies of the safety of antimalarials in pregnancy and lactation are few. The only recommended medication used for radical treatment of P.vivax is primaquine. The 2010 WHO malaria guidelines recommend its use in all patients with P.vivax infection in areas of low transmission, in the absence of contraindications. Primaquine is contraindicated in pregnancy. The postpartum period presents a key opportunity to definitively treat women who suffer multiple malaria relapses during pregnancy. The 2010 WHO malaria treatment guidelines allow for primaquine use during lactation but there are no studies to date quantifying primaquine excretion in breast milk and the dose that breastfed infants would be exposed to is unknown. The investigators propose to study the pharmacokinetics of primaquine in maternal and infant plasma and in breast milk during a 14 day radical treatment of P.vivax.

Rationale

The global burden of malaria is great, with approximately 1-2 million deaths each year and many times that number of productive days lost to illness. Plasmodium vivax is the most prevalent malarial species, resulting in 132-391 million clinical infections each year and 80-90% of malaria in Asia, the Middle East, and the Western Pacific. Despite its prevalence, P.vivax has not been a focus of research until recently, and its effects and optimal treatments are still not fully understood. Though infrequently a fatal infection, P.vivax causes high levels of morbidity due to the chronic nature of the infection. Because of dormant liver stages (hypnozoites), illness can continue to recur for years, even after effective treatment has eliminated the parasites from the blood. In settings where there are hopes for malarial eradication, this means infected persons continue to be hosts even if vector-borne transmission is temporarily interrupted, and could potentially start a new cycle of transmission with each relapse. Each of these relapses causes a significant amount of morbidity and a small mortality risk for those infected.

These burdens are magnified during pregnancy when women experience relative immune suppression and can experience relapses every 4-8 weeks. P.vivax malaria in pregnancy is associated with low birth weight and anaemia; thrombocytopaenia; increased risk of fetal loss, premature delivery, neonatal and infant mortality; and, in some areas, risk for congenital malaria (a severe, sepsis-like illness). In Southeast Asia, where the investigators propose to conduct our study, the majority of cases of congenital malaria are from vivax infection. These women may have some respite during the postpartum period, with relapses spaced further apart, but frequently relapse again in subsequent pregnancies. New pregnancies during the end of lactation are common in many malaria endemic areas, including our setting, making definitive treatment of vivax infections in these women very challenging in the absence of data about the safety of primaquine for the breastfeeding infant.

Though the anti-malarial pharmacopeia has expanded over the past decade, primaquine remains the only definitive treatment for the hypnozoite forms of Plasmodium vivax and ovale. First synthesized in 1946, a 14 day treatment eradicates the parasites from the liver. However, this medication has been associated with a risk for methemoglobinemia, and acute intravascular haemolysis in glucose-6-phosphate-dehydrogenase (G6PD) deficient hosts (common in malaria-endemic areas). The elevations in methemoglobin are generally modest and asymptomatic, but occasionally significant methemoglobinemia can cause cyanosis and shortness of breath requiring discontinuation of the medication. Primaquine is not considered safe in pregnancy because of the possible risk of haemolysis and methaemoglobin in the fetus. The most recent WHO malaria guidelines (2010) have conflicting information about the its use during lactation. They cite breastfeeding as a contraindication for primaquine administration for P. falciparum malaria, but permit the use of primaquine for P. vivax during lactation if the breast fed infant is not G6PD deficient. No studies have ever been done in lactating women to determine the safety of primaquine in breastfeeding or the optimal time of administration, however, the relaxation of guidelines in infancy suggest potential for its safe use in lactation. Some authors note that primaquine's once daily dosing might allow for safe breastfeeding if the mother pumps the milk at the time when peak milk concentrations are expected and discards that milk.

Some inferences about the expected behavior of primaquine in lactation can be drawn from its known pharmacologic properties. Primaquine pharmacokinetics have been well characterized in healthy subjects and malaria patients after single and multiple oral dosing. Peak concentrations are reached within 2-3 hours after dosing and the plasma elimination half-life is ~7 hours. It is extensively distributed in the tissue and largely metabolized to inert carboxyprimaquine, the major plasma metabolite, which undergoes further biotransformation to unknown metabolites that are probably more toxic than the parent compound. The identification of other metabolites in humans has been difficult to pursue because the expected aminophenol metabolites are unstable. Until recently, techniques to separate positive and negative enantiomers for primaquine and carboxyprimaquine have not been possible, again obscuring the toxic and therapeutic mechanisms of the drug.

Primaquine has limited oral bioavailability and adult plasma concentrations are generally low, making dangerously high concentrations in maternal milk unlikely from a theoretical standpoint. However, recent data suggests that a previously unrecognized sex difference exists in the pharmacokinetics of the medication in men and women, with women accumulating higher drug concentrations than men. Since side effects of primaquine appear to be dose-related, this finding could be significant. The time to maximum concentration is about 2-3 hrs (longer for women than for men) and the investigators would expect to see a short lag in reaching peak breast milk concentrations. Primaquine has a low molecular weight (259) and slightly basic pH making it more likely to transfer into the breast milk.

Literature on medication pharmacokinetics in breast milk is sparse but has begun to capture the interest of researchers and human rights activists who note that women are often systematically excluded from medical research by virtue of pregnant or lactating status. As a result, during these two states the pharmacokinetic properties of drugs remain poorly understood, and much of our clinical therapeutic approaches are based on consensus and conjecture. No pharmacokinetic studies have been done to measure primaquine excretion in breast milk. A few studies have been done of other antimalarials during lactation and have shown low levels of drug in breast milk during treatment. The frequent venous sampling necessary for pharmacokinetic research is not ideal for participants, especially in pediatric populations. Recent efforts have been made to evaluate the usefulness of capillary or saliva samples as alternative sampling measures.

ELIGIBILITY:
Inclusion Criteria:

* Lactating women aged 18 years and older who are breast feeding one infant aged more than 28 days.
* G6PD normal
* History of proven P.vivax malaria that has not been treated with primaquine
* Willingness and ability to comply with the study protocol for the duration of the trial
* Written informed consent provided

Exclusion Criteria:

* Known hypersensitivity to primaquine, defined as history of erythroderma/other severe cutaneous reaction, angioedema or anaphylaxis
* Glucose-6-phosphate-dehydrogenase (G6PD) deficiency in mother
* Glucose-6-phosphate-dehydrogenase (G6PD) deficiency in infant
* Pregnancy (urine test for HCG to be performed on any woman of child bearing age unless menstruating)
* Blood smear positive for malaria at the time of enrolment
* Presence of intercurrent illness or any condition which in the judgement of the investigator would place the patient at undue risk or interfere with the results of the study
* Hematocrit (HCT) <25% in the mother or <33% in the infant
* Use of medications other than antipyretics in the past 7 days or Chloroquine in the past 2 months.
* Use of primaquine since most recent malaria episode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameters of Primaquine and Carboxyprimaquine in breast milk. Area Under Curve (AUC) | 13 Days. Time Frame: predose, 0,1,2,3,4,6,8,12,24,72 hours; Day 7, Day 13 post-dose
  Primaquine and carboxyprimaquine pharmacokinetic parameters to day 13 in breast milk of lactating women treated with primaquine for radical treatment of P.vivax.

SECONDARY OUTCOMES:
Pharmacokinetics Parameters of Primaquine and Carboxyprimaquine in blood. Area Under Curve (AUC). | 13 Days. Time Frame: predose, 0,1,2,3,4,6,8,12,24,72 hours; Day 7, Day 13 post-dose
  Primaquine and carboxyprimaquine pharmacokinetic parameters to day 13 in the blood of lactating women and their breastfed infants
Concentration of Primaquine in saliva and urine. Area Under Curve (AUC). | 13 Days. Time Frame: predose, 0,1,2,3,4,6,8,12,24,72 hours; Day 7, Day 13 post-dose
  Primaquine concentration in saliva and urine.
Primaquine dosage in infant - the relative infant dose. Area Under Curve (AUC). | 13 Days. Time Frame: predose, 0,1,2,3,4,6,8,12,24,72 hours; Day 7, Day 13 post-dose
  Relative infant dose of Primaquine.
Assessment of adverse events during primaquine administration | 63 days
  Adverse events in mothers and infants during treatment. Number of Participants with Adverse Events as a Measure of Safety and Tolerability.
Hematocrit levels in mother and child | 63 days
  Changes in maternal and infant hematocrit to day 63.

CONTACTS AND LOCATIONS:
Overall Officials: Rose McGready, MD, Principal Investigator — University of Oxford
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

REFERENCES:
- [Derived] Wattanakul T, Gilder ME, McGready R, Hanpithakpong W, Day NPJ, White NJ, Nosten F, Tarning J, Hoglund RM. Population pharmacokinetic modelling of primaquine exposures in lactating women and breastfed infants. Nat Commun. 2024 May 8;15(1):3851. doi: 10.1038/s41467-024-47908-y. PMID 38719803
- [Derived] Gilder ME, Hanpithakphong W, Hoglund RM, Tarning J, Win HH, Hilda N, Chu CS, Bancone G, Carrara VI, Singhasivanon P, White NJ, Nosten F, McGready R. Primaquine Pharmacokinetics in Lactating Women and Breastfed Infant Exposures. Clin Infect Dis. 2018 Sep 14;67(7):1000-1007. doi: 10.1093/cid/ciy235. PMID 29590311